CLINICAL TRIAL: NCT00449020
Title: Carboplatin and Irinotecan Concomitantly With Radiation Therapy Followed by Consolidation Chemotherapy With Docetaxel for Locally Advanced Non-Small Cell Lung Cancer (GIA 12177).
Brief Title: Carboplatin, Irinotecan, and Radiation Therapy Followed By Docetaxel in Treating Patients With Newly Diagnosed Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030244; SCCC-2003049 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20051708 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Docetaxel; Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Carboplatin — CARBOPLATIN (AUC=2) IV in 250 cc NS over 30 minutes, weekly for seven weeks (Days #1, #8, #15, #22, #29, #36 and #43) along with radiation.
Drug: Docetaxel — DOCETAXEL 75 mg/m2 IV over one hour every three weeks for 3 cycles.
Drug: irinotecan hydrochloride — IRINOTECAN 30 mg/m2 IV over 90 minutes weekly for seven weeks (Days #1, #8, #15, #22, #29, #36 and #43) along with radiation.
Radiation: radiation therapy — Radiotherapy will start on the first day of scheduled chemotherapy. The daily administered dose will be 1.8 Gy, 5 days a week for 4.4 weeks, 22 fractions, ( 39.6 Gy) to the primary tumor and mediastinum (primary planning target volume: PPTV). After 39.6 Gy, the same targets will be treated by oblique fields at 1.8 GY for 3 fxs to a toal dose of 45 GY. Thereafter, the primary tumor and involved nodal metastasis (secondary planning target volume SPTV) will be boosted at 2 Gy per day to 18 Gy in 9 fractions. The total dose will be 63 Gy in 35 fractions over seven weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, irinotecan, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin and irinotecan together with radiation therapy followed by docetaxel works in treating patients with newly diagnosed stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with newly diagnosed stage IIIA or IIIB non-small cell lung cancer treated with concurrent carboplatin, irinotecan hydrochloride, and radiotherapy followed by consolidation docetaxel.

Secondary

* Evaluate the safety, toxicity, and complications of this regimen in these patients.
* Evaluate the median survival, 1-year and 2-year survival, and time to tumor progression in these patients.

OUTLINE:

* Chemoradiotherapy: Patients receive carboplatin IV over 30 minutes followed by irinotecan hydrochloride IV over 90 minutes on day 1. Patients also undergo radiotherapy once daily on days 1-5. Treatment repeats weekly for up to 7 courses in the absence of disease progression or unacceptable toxicity.
* Consolidation chemotherapy: Beginning 3-4 weeks after completion of chemoradiotherapy, patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIA or IIIB disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques or > 10 mm by spiral CT scan
* No clinically significant malignant pleural or pericardial effusion (i.e., stage IIIB wet disease)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin normal
* Alkaline phosphatase (AP), AST, and ALT meeting 1 of the following criteria:

  * AP normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal
* Creatinine < 2.0 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No New York Heart Association class III-IV heart disease
* No history of serious cardiac disease not adequately controlled
* No documented myocardial infarction within the past 6 months
* No congestive heart failure
* No unstable angina
* No clinically significant arrhythmia
* No history of severe hypersensitivity reaction to drugs formulated with polysorbate 80
* No peripheral neuropathy > grade 1
* No other malignancy within the past 5 years other than skin cancer

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior major surgery
* No prior systemic chemotherapy, thoracic radiotherapy, or surgical resection for NSCLC

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-01; Primary Completion 2007-05 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Response (complete response, partial response, overall response) as measured by RECIST criteria prior to course 1 and within 1 month after completion of course 3 of consolidation chemotherapy | 5.25 years

SECONDARY OUTCOMES:
Toxicity/safety profile as measured by NCI CTCAE v 3.0 | 5.25 years
Median survival | 5.25 years
1-year survival | 5.25 years
2-year survival | 5.25 years
Time to disease progression | 5.25 years

CONTACTS AND LOCATIONS:
Overall Officials: Luis E. Raez, MD, FACP, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

REFERENCES:
- [Result] Bastos BR, Hatoum GF, Walker GR, Tolba K, Takita C, Gomez J, Santos ES, Lopes G, Raez LE. Efficacy and toxicity of chemoradiotherapy with carboplatin and irinotecan followed by consolidation docetaxel for unresectable stage III non-small cell lung cancer. J Thorac Oncol. 2010 Apr;5(4):533-9. doi: 10.1097/JTO.0b013e3181ce3e00. PMID 20357618